CLINICAL TRIAL: NCT04140526
Title: Safety, Pharmacokinetics (PK), and Efficacy of ONC-392 as a Single Agent and in Combination With Pembrolizumab in Advanced Solid Tumors and NSCLC: An Open Label Phase IA/IB Study. Preserve CTLA4 Checkpoint Function (PRESERVE-001)
Brief Title: Safety, PK and Efficacy of ONC-392 in Monotherapy and in Combination of Anti-PD-1 in Advanced Solid Tumors and NSCLC
Acronym: PRESERVE-001
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-392-001; 4R44CA250824-02 (NIH); 20193108 (Other: WIRB)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer; Advanced Solid Tumor; Metastatic Melanoma; Metastatic Head and Neck Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Colorectal Cancer; Sarcomas; Metastatic Prostate Cancer; Ovarian Cancer; Small Cell Lung Cancer; Metastatic Breast Cancer; Pancreas Cancer; Gastric Cancer; Esophageal Cancer; Gastroesophageal Junction Adenocarcinoma; Cervical Cancer; Adenoid Cystic Carcinoma; Salivary Gland Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Colorectal Neoplasms; Sarcoma; Prostatic Neoplasms; Ovarian Neoplasms; Small Cell Lung Carcinoma; Breast Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Adenoid Cystic; Salivary Gland Neoplasms; Carcinoma, Transitional Cell | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ONC-392 Treatment as single agent (Experimental): The Part A study will test ONC-392 intravenous (IV) infusion up to five predefined dose levels from 0.1 mg/kg to 10 mg/kg ONC-392 as monotherapy every 21 days (Q3W). The Part A study will determine the maximal tolerable dose (MTD) and the recommended Phase 2 dose in monotherapy (RP2D-M).
  In Part C, Arms A-C, I-N monotherapy expansion cohorts will further assess the safety and efficacy of ONC-392 in different dose levels as monotherapy in pancreatic cancer, triple negative breast cancer, non small cell lung cancer with driver mutations, PD-1 resistant non small cell lung cancer, PD-1 resistant melanoma, head and neck cancer, ovarian cancer, renal cell carcinoma and other solid tumors.
  Part D is a Phase II study on recurrent and/or metastatic adenoid cystic carcinoma.
  Interventions: Drug: ONC-392
- ONC-392 in combination with pembrolizumab (Experimental): The Part B1 study will test ONC-392 intravenous (IV) infusion, Q3W, in combination with fixed dose of pembrolizumab. The dose for pembrolizumab will be fixed at 200mg/cycle dosed every 21 days (Q3W).
  The Part B1 will start at one level below RP2D-M dose for ONC-392 and 200mg of pembrolizumab. When 2 DLTs occur before 6 patients are enrolled, the ONC-392 dose will be decreased to the next dose level until ≤ 1/6 patients treated at that dose develops a DLT. This dose level will be designated RP2D-C.
  In Part C, the expansion cohorts Arm D to G will assess the safety and efficacy of ONC-392 in different dose levels and Pembrolizumab combination therapy in non small cell lung cancer, and metastatic melanoma.
  Interventions: Drug: ONC-392; Drug: Pembrolizumab
- ONC-392 and docetaxel (Experimental): Part E Arm O will test ONC-392 in combination with docetaxel, IV infusion, Q3W, in PD-1 resistant NSCLC patients.
  Interventions: Drug: ONC-392; Drug: Docetaxel

INTERVENTIONS:
Drug: ONC-392 — ONC-392 will be given by intravenous infusion, once every 21 days (Q3W). In Part C Arm M and in Part D, ONC-392 will be given Q4W.
  Other Names: A humanized anti-CTLA4 IgG1 monoclonal antibody made by OncoC4, Inc.
Drug: Pembrolizumab — Pembrolizumab will be given intravenous (IV) infusion at 200 mg/cycle, once every 21 days (Q3W).
  Other Names: Keytruda; MK3475
  Arms: ONC-392 in combination with pembrolizumab
Drug: Docetaxel — Docetaxel will be given intravenous (IV) infusion at 75 mg/m2, once every 21 days (Q3W).
  Other Names: Taxotere, Docefrez
  Arms: ONC-392 and docetaxel

SUMMARY:
This is a First-in-Human Phase IA/IB/II open label dose escalation study of intravenous (IV) administration of ONC-392, a humanized anti-CTLA4 IgG1 monoclonal antibody, as single agent and in combination with pembrolizumab in participants with advanced or metastatic solid tumors and non-small cell lung cancers.

DETAILED DESCRIPTION:
Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), also known as CD152 (cluster of differentiation 152), is a cell surface protein receptor that interacts with B7-1 (CD80) and B7-2 (CD86) to ensure proper function of regulatory T cells and protect host against autoinflammatory diseases. Anti-CTLA-4 monoclonal antibodies (mAbs) have demonstrated strong and broad cancer immunotherapeutic effects (CITE) in a variety of preclinical models and are used clinically both as monotherapy and as part of combination therapy with Nivolumab (anti-PD-1). However, CTLA-4 monotherapy has more immunotherapy-related adverse effects (irAEs) than anti-PD-1/PD-L1 therapy. In addition, the rate of severe irAE (Grades 3 and 4) reached 55% in melanoma patients receiving combination of Ipilimumab and Nivolumab. The strong irAEs further limit the doses tolerated by cancer patients. Nevertheless, combination with anti-PD-1 resulted in significantly improved response rates and patient survival in multiple types of cancer. Furthermore, anti-CTLA-4 antibodies induce long-lasting immunity in cancer patients. Therefore, CTLA-4 remains an important immunotherapy target, but major challenges remain in improving both safety and efficacy of anti-CTLA-4 mAbs.

ONC-392 is a highly selective, humanized monoclonal IgG1-kappa isotype antibody against CTLA-4. The parental clone was identified through in vivo screening in humanized CTLA-4 mouse model for high anti-tumor efficacy and low autoimmune toxicity. We have recently demonstrated that ONC-392 is dissociation from CTLA-4 under low pH to allow its escape from lysosomal degradation and recycle to cell surface. We have provided several lines of evidence for the notion that a pH-sensitive antibody ONC-392 is not only safer but also more effective in Treg depletion and tumor rejection than the Ipilimumab, which is pH-insensitive. First, by preserving CTLA-4 on the cell surface, Onc-392 leaves higher ligand density for better ADCC.

Second, Onc-392 is more efficient in Treg depletion in tumor microenvironment. Third, Onc-392 is significantly more potent in inducing rejection of large tumors.

The study consists of four parts:

(1) The Part A study is a dose-finding rapid titration, Phase I trial of ONC-392 as a single agent in patients with advanced or metastatic solid tumors with various histology. The aim of this trial is to define the recommended Phase II dose for ONC-392 monotherapy (RP2D-M). (2) The Part B study is a dose-finding phase with ONC-392 in combination with a standard dose of 200 mg pembrolizumab in patients with advanced or metastatic solid tumors.

(3) The Part C consists of different expansion arms.

1. Arm A: Pancreatic Cancer Cohort, ONC-392 monotherapy, will enroll advanced/metastatic pancreatic cancer patients who have progressive disease after first and second lines of systemic treatment.
2. Arm B: TNBC Cohort, ONC-392 monotherapy, will enroll advanced/metastatic TNBC patients who have progressive disease after prior systemic treatments, including checkpoint inhibitor immunotherapy.
3. Arm C: NSCLC Mono Cohort 1, ONC-392 monotherapy, will enroll advanced/metastatic NSCLC patients with EGFR or ALK mutations who have progressive disease after prior systemic treatments, including targeted therapy or checkpoint inhibitors.
4. Arm D: NSCLC IO Naïve Cohort, ONC-392/Pembrolizumab combination therapy, will enroll advanced/metastatic NSCLC cancer patients who are treatment naïve, or anti PD (L)1 immunotherapy naïve and PD-L1-positive (PD L1 TPS ≥ 1%).
5. Arm E: NSCLC IO R/R Cohort, ONC-392/Pembrolizumab combination therapy, will enroll advanced/metastatic NSCLC cancer patients who are R/R to prior anti-PD-(L)1 immunotherapy regardless of PD-L1 status.
6. Arm F: Melanoma IO Naïve Cohort, ONC-392/Pembrolizumab combination therapy, will enroll advanced/metastatic Melanoma patients who are treatment naïve, or checkpoint inhibitor immunotherapy naive. Prior systemic chemotherapy or targeted therapy are allowed.
7. Arm G: Melanoma IO R/R Cohort, ONC-392/Pembrolizumab combination therapy, will enroll advanced/metastatic melanoma patients who are R/R to anti-PD-(L)1 immunotherapy.
8. Arm I: NSCLC Mono Cohort 2, ONC-392 monotherapy, will enroll advanced/metastatic NSCLC patients without EGFR or ALK mutations who have progressive disease after prior systemic treatments, including chemotherapy or checkpoint inhibitors. Patient must have anti-PD-(L)1 treatment, either alone or in combination, as last treatment before enrollment. Prior anti-CTLA-4 treatment is allowed.
9. Arm J: Melanoma Mono Cohort, ONC-392 monotherapy, will enroll advanced/metastatic melanoma patients who are R/R to anti-PD-(L)1 immunotherapy.
10. Arm K: Head and Neck Squamous Cell Carcinoma (HNSCC), ONC-392 monotherapy, will enroll advanced/metastatic HNSCC patients with or without positive HPV who have progressive disease after prior systemic treatments, including chemotherapy or checkpoint inhibitors. Patient must have anti-PD-(L)1 treatment, either alone or in combination, as last treatment before enrollment.
11. Arm L: Ovarian Cancer, ONC-392 monotherapy, will enroll patients with advanced/metastatic ovarian cancer who have progressive disease after prior systemic treatments, including chemotherapy, targeted therapy or checkpoint inhibitors.
12. Arm M: Solid Tumors, ONC-392 monotherapy, will enroll patients with advanced/metastatic solid tumors who are not eligible for Arm A-C or H-L, who have progressive disease after prior systemic treatments, including chemotherapy, targeted therapy or checkpoint inhibitors.
13. Arm N: Renal Cell Carcinoma, ONC-392 monotherapy, will enroll advanced/metastatic RCC patients who are R/R to anti-PD-(L)1 immunotherapy.

(4) Part D is a Phase II study in recurrent and/or metastatic adenoid cystic carcinoma with ONC-392 monotherapy.

(5) Part E Arm O will test ONC-392 in combination with docetaxel in PD-1 resistant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. . Patients must have a histological or cytological diagnosis of NSCLC or any other type of carcinoma or sarcomas, progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy.

   1. In the Part A Phase I dose escalation study of ONC-392 monotherapy, patients with advanced/metastatic solid tumors of any histology are eligible for participation.

      Please note: tumor types of primary interest in this study are malignant melanoma, renal cell carcinoma, hepatocellular carcinoma, non-small cell lung cancer, head and neck carcinoma, gastric carcinoma, ovarian carcinoma, colorectal cancer, any type of sarcoma.
   2. In Part B dose finding of the ONC-392 plus pembrolizumab combination, patients with advanced/metastatic solid tumors of any histology that Pembrolizumab has been approval as standard of care are eligible for participation.
   3. In Part C, patients with pancreatic cancer, triple negative breast cancer, non small cell lung cancer, melanoma, Head and Neck cancer, ovarian cancer, and other solid tumors are eligible.
   4. In Part D, patients with recurrent and/or metastatic adenoid cystic carcinoma with disease progression within 12 months are eligible.
   5. Patients must have RECIST V1.1 Measurable disease:
2. Patient is male or female and >18 years of age on day of signing informed consent.
3. Patient must have a performance status of 0 or 1 on the ECOG Performance Scale
4. Patient must have adequate organ function as indicated by the following laboratory values:

   Hematological: Absolute neutrophil count (ANC) ≥1,500 /mcL; Plateletsa ≥100,000 / mcL; Hemoglobin ≥9 g/dL or ≥5.6 mmol/L- without qualifications; Renal: Serum creatinine ≤1.5 X upper limit of normal (ULN); Hepatic: Serum total bilirubin ≤1.5 X ULN; OR Direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 ULN; AST (SGOT) and ALT (SGPT) ≤2.5 X ULN, OR ≤5 X ULN for patients with active liver metastases Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN
5. Patient has voluntarily agreed to participate by giving written informed consent.
6. Female patient of childbearing potential has a negative urine or serum pregnancy test.
7. Female and Male patients must agree to use adequate methods of contraception starting with the first dose of study drug through 90 days after the last dose of study therapy.

Exclusion Criteria:

A patient meeting any of the following criteria is not eligible to participate in this study:

1. Patients who have not recovered to CTCAE ≤ 1 from the AE due to cancer therapeutics. The washout period for cancer therapeutic drugs (such as chemotherapy, radioactive, or targeted therapy) is 21 days, and for antibody drug 28 days.
2. Patients who are currently enrolled in a clinical trial of an investigational agent or device.
3. Patients who are on chronic systemic steroid therapy at doses >10 mg/day
4. Patients who have active symptomatic brain metastasis or leptomeningeal metastasis.
5. Patients who have an active infection requiring systemic IV therapy within 14 days of prior to administration of ONC-392 or combined ONC-392 and Pembrolizumab.
6. Patients who have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
7. Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. Patients who are pregnant or breastfeeding.
9. For the Part B and Part C Arm D to G, the patients that are deemed to be not suitable for Pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) in monotherapy | 21 days
  The number of subjects who have dose limiting toxicity during the first cycle of study drug, ONC-392, administration.
Maximal tolerable dose (MTD) in monotherapy | 21 days
  The study drug, ONC-392, dose level that has two out of six subjects who have dose limiting toxicity.
Recommended Phase II Dose (RP2D) | 21 days
  The study drug, ONC-392, dose level that is one level below MTD, or an intermediate dose level that below MTD and pre-specified in protocol. This dose level will be the RP2D for monotherapy.
Rate of treatment related adverse events (TRAE) according to CTCAE v5.0 | One year
  The safety profile will be presented as tabulated TRAE.

SECONDARY OUTCOMES:
The serum half life of the study drug, ONC-392, in monotherapy. | 12 weeks
  To determine the drug concentration in serum samples that are taken in various timepoints during the treatment in order to calculate drug half life.
The serum half life of the study drug, ONC-392, in combination therapy with Pembrolizumab. | 12 weeks
  To determine the drug concentration in serum samples that are taken in various timepoints during the treatment in order to calculate drug half life.
Objective Response Rate (ORR) | 1 year
  To determine the objective response rate based on RECIST v1.1.
Progression Free Survival (PFS) | 1 year
  To determine the progression free survival based on RECIST 1.1 and iRECIST.
Overall Survival (OS) | 1 year
  To determine the overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Tianhong Li, MD, Principal Investigator — University of California, Davis
Locations (37):
- United States (33):
  - Highlands Oncology Group, Springdale, Arkansas
  - University of California at Davis, Davis, California
  - The Oncology Institute of Hope and Innovation, Downey, California
  - City of Hope Cancer Center, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - Nuvance Health, Norwalk, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Atlantis, Florida
  - University of Florida Health Cancer Center, Gainesville, Florida
  - Ocala Oncology Florida Cancer Affiliates, Ocala, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Norton Health, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Atlantic Healthcare System, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University James Cancer Center, Columbus, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Pennsylvania Cancer Specialists & Research Institute (Formerly Gettysburg Cancer Center), Gettysburg, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Tennessee Oncology Chattanooga Memorial Plaza, Chattanooga, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT/Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Tasman Oncology Research, Southport, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Du X, Liu M, Tang F, Zhang P, Ai C, Fields JK, Sundberg EJ, Latinovic OS, Devenport M, Zheng P, Liu Y. Hijacking antibody-induced CTLA-4 lysosomal degradation for safer and more effective cancer immunotherapy. Cell Res. 2019 Aug;29(8):609-627. doi: 10.1038/s41422-019-0184-1. Epub 2019 Jul 2. PMID 31267017
- [Background] Du X, Tang F, Liu M, Su J, Zhang Y, Wu W, Devenport M, Lazarski CA, Zhang P, Wang X, Ye P, Wang C, Hwang E, Zhu T, Xu T, Zheng P, Liu Y. A reappraisal of CTLA-4 checkpoint blockade in cancer immunotherapy. Cell Res. 2018 Apr;28(4):416-432. doi: 10.1038/s41422-018-0011-0. Epub 2018 Feb 22. PMID 29472691
- [Background] Du X, Liu M, Su J, Zhang P, Tang F, Ye P, Devenport M, Wang X, Zhang Y, Liu Y, Zheng P. Uncoupling therapeutic from immunotherapy-related adverse effects for safer and effective anti-CTLA-4 antibodies in CTLA4 humanized mice. Cell Res. 2018 Apr;28(4):433-447. doi: 10.1038/s41422-018-0012-z. Epub 2018 Feb 20. PMID 29463898
- [Background] May KF Jr, Roychowdhury S, Bhatt D, Kocak E, Bai XF, Liu JQ, Ferketich AK, Martin EW Jr, Caligiuri MA, Zheng P, Liu Y. Anti-human CTLA-4 monoclonal antibody promotes T-cell expansion and immunity in a hu-PBL-SCID model: a new method for preclinical screening of costimulatory monoclonal antibodies. Blood. 2005 Feb 1;105(3):1114-20. doi: 10.1182/blood-2004-07-2561. Epub 2004 Oct 14. PMID 15486062
- [Background] Lute KD, May KF Jr, Lu P, Zhang H, Kocak E, Mosinger B, Wolford C, Phillips G, Caligiuri MA, Zheng P, Liu Y. Human CTLA4 knock-in mice unravel the quantitative link between tumor immunity and autoimmunity induced by anti-CTLA-4 antibodies. Blood. 2005 Nov 1;106(9):3127-33. doi: 10.1182/blood-2005-06-2298. Epub 2005 Jul 21. PMID 16037385
- [Background] Liu Y, Zheng P. Preserving the CTLA-4 Checkpoint for Safer and More Effective Cancer Immunotherapy. Trends Pharmacol Sci. 2020 Jan;41(1):4-12. doi: 10.1016/j.tips.2019.11.003. Epub 2019 Dec 10. PMID 31836191
- [Background] Li T, Tang M, Kelly, K, Chen HA, Joo S, Khan I, Do N, Touomou R, Chen D, Liu Y, Zheng P. 949 First-in-human study of the first acid pH-sensitive and recycling CTLA-4 antibody that preserves the immune tolerance checkpoint to avoid immunotherapy-related adverse events in cancer patients. Journal for ImmunoTherapy of Cancer, 2021. 9(Suppl 2): p. A998-A998. doi: 10.1136/jitc-2021-SITC2021.949
- [Background] Hu-Lieskovan S, He K, Tang M, Chen D, Liu Y, Zheng P, Li T. 594 Dose escalation of next generation anti-CTLA-4 antibody ONC-392 in combination with fixed dose of pembrolizumab in patients with advanced solid tumors. Journal for ImmunoTherapy of Cancer, 2022. 10(Suppl 2): p. A622-A622. doi: 10.1136/jitc-2022-SITC2022.0594
- [Background] He K, Carbone DP, McKean M, Balaraman R, Shah S, Arrowsmith E, Peguero JA, Joshi R, He AR, Milillo A, Hamm JT, Goldstein MG, Li Z, Liu Y, Zheng P, Li T. Safety and clinical activity of target-preserving anti-CTLA-4 antibody ONC-392 as monotherapy in NSCLC patients who progressed on PD(L)1-targeted immunotherapy. Journal of Clinical Oncology, 2023. 41(16_suppl): p. 9024-9024. doi: 10.1200/JCO.2023.41.16_suppl.9024
- [Background] He K, McKean M, Balaraman R, Shah S, Arrowsmith E, Peguero JA, Hamm JT, He AR, Spira AI, Milillo-Naraine A, Joshi R, Goldstein MG, Carbone DP, Tang M, Hu-Lieskovan S, Li Z, Chen D, Chou HY, Yang J, Liu Y, Zheng P, Li T. 599 Single-agent safety and activities of target-preserving anti-CTLA-4 antibody gotistobart (ONC-392/BNT316) in PD-(L)1 resistant metastatic NSCLC and population PK analysis in patients with solid tumors. Journal for ImmunoTherapy of Cancer, 2023. 11(Suppl 1): p. A682-A682. doi: 10.1136/jitc-2023-SITC2023.0599